CLINICAL TRIAL: NCT04438382
Title: Optimizing Immunosuppression for Steroid-Refractory Anti-PD-1/PD-L1 Pneumonitis
Brief Title: Infliximab and Intravenous Immunoglobulin Therapy in Treating Patients With Steroid-Refractory Pneumonitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAQ172; NCI-2018-02825 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ172 (Other: ECOG-ACRIN Cancer Research Group); EAQ172 (Other: DCP); EAQ172 (Other: CTEP); UG1CA189828 (NIH)
Record Dates: First submitted 2020-06-09; First posted 2020-06-18 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Steroid-Refractory Pneumonitis
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Infliximab; gamma-Globulins; Immunoglobulins; Immunoglobulins, Intravenous; Prednisone; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (infliximab) (Experimental): Patients receive infliximab IV on day 1 followed by prednisone taper IV or PO for 4-6 weeks in the absence of disease progression or unacceptable toxicity. Patients may receive an additional dose of infliximab IV on day 14 at the discretion of the treating physician.
  Interventions: Biological: Infliximab; Drug: Prednisone; Drug: Methylprednisolone
- Arm B (intravenous immunoglobulin therapy) (Experimental): Patients receive intravenous immunoglobulin therapy IV over 2-5 days per institutional guidelines followed by prednisone taper IV or PO for 4-6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Intravenous Immunoglobulin Therapy; Drug: Prednisone; Drug: Methylprednisolone

INTERVENTIONS:
Biological: Infliximab — Given IV
  Other Names: Remicade
  Arms: Arm A (infliximab)
Biological: Intravenous Immunoglobulin Therapy — Given IV
  Other Names: Gamma Globulin; Gamma Globulin Therapy; Immune Globulin; Immune Globulin Therapy; Intravenous Immunoglobulin; IVIG
  Arms: Arm B (intravenous immunoglobulin therapy)
Drug: Prednisone — Given IV or PO
  Other Names: Deltasone; Orasone; Meticorten; Panasol-S; Liquid-Pred
Drug: Methylprednisolone — Given IV or PO
  Other Names: Methylprednisolone sodium succinate (Solu-Medrol); methylprednisolone acetate (Depo-Medrol); Methylprednisolone (Medrol)

SUMMARY:
This phase II trial studies how well infliximab and intravenous immunoglobulin therapy work in treating patients with pneumonitis that does not respond to steroid treatment. Immunotherapy with monoclonal antibodies such as, infliximab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Intravenous immunoglobulin therapy may improve pneumonitis. It is not yet known whether giving infliximab and intravenous immunoglobulin therapy will work better in treating patients with pneumonitis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess pneumonitis response to additional immunosuppression (infliximab or intravenous immunoglobulin therapy [IVIG]) in patients with steroid-refractory pneumonitis at 28-days.

SECONDARY OBJECTIVES:

I. To assess functional parameters of steroid-refractory pneumonitis at day 1, 14-days and 28-days after day 1 of receipt of additional immunosuppression (infliximab or IVIG).

II. To assess radiologic parameters of steroid-refractory pneumonitis at day 1, 14-days and 28-days after day 1 of receipt of additional immunosuppression (infliximab or IVIG).

III. To assess patient-reported outcomes of steroid-refractory pneumonitis at day 1, 14-days and 28-days after day 1 of receipt of additional immunosuppression (infliximab or IVIG).

IV. To assess death after additional immunosuppression. V. To assess the rate of infections in the 28-day period after additional immunosuppression.

EXPLORATORY OBJECTIVES:

I. To examine lung tissue, bronchoalveolar lavage (BAL) and serial blood samples in patients who develop steroid-refractory pneumonitis.

II. To examine associations between BAL phenotypes and pneumonitis response, functional and radiologic parameters of pneumonitis.

III. To evaluate associations between pneumonitis and autoantibodies, T-cell expansion, and baseline cytokines in the blood.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive infliximab intravenously (IV) on day 1 followed by prednisone taper IV or orally (PO) for 4-6 weeks in the absence of disease progression or unacceptable toxicity. Patients may receive an additional dose of infliximab IV on day 14 at the discretion of the treating physician.

ARM B: Patients receive intravenous immunoglobulin therapy IV over 2-5 days per institutional guidelines followed by prednisone taper IV or PO for 4-6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28, 42 and 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be English-speaking and be able to provide informed consent
* Patient must be willing and able to undergo arterial blood gas assessment as per the treating investigator. Patient must not have contraindication for arterial blood gas assessment
* Women must not be pregnant or breast-feeding due to the potential risk to the fetus of infliximab or IVIG. All females of childbearing potential must have a blood test or urine test within 14 days prior to randomization to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method(s) of contraception or to abstain from sexual intercourse for a minimum of 56 days (the duration of their participation in the study)
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Patient may have received any number of lines of prior systemic therapy
* Patient may have any solid tumor or hematologic malignancy is eligible
* Patient must have received treatment with an anti-PD-1/PD-L1 agent either alone or in combination with another anti-cancer agent, as their most recent therapy prior to development of pneumonitis
* Patient must have steroid-refractory pneumonitis defined as:

  * Grade 2 pneumonitis that has not clinically improved by a Common Terminology Criteria for Adverse Events (CTCAE) grade in greater than 72 hours or maximum of 14 days or
  * Grade 3 or higher pneumonitis that has not clinically improved by a CTCAE grade in greater than 48 hours or maximum of 14 days with high dose corticosteroids (methylprednisolone or prednisone 1-4 mg/kg/equivalent) as their most recent treatment for pneumonitis, as determined by the treating investigator
* Patient may have received anti-PD-1/PD-L1 therapy as standard-of-care or part of a clinical trial
* Patient must have had pathogen-negative infectious diagnostic evaluation within 14 days prior to randomization, and at a minimum these should include: blood culture, urine culture, sputum culture, and viral panel: rapid flu, respiratory syncytial virus (RSV), herpes simplex virus (HSV). Empiric antibiotics for culture negative infections are not an exclusion for study entry
* Patient must have had a pathogen-negative bronchoscopic assessment of BAL fluid within 14 days prior to randomization. A minimum assessment for pathogens on BAL must include: gram stain, fungal panel, viral panel
* Patient must have a negative tuberculosis assessment (TB spot test, quantiferon gold or tuberculin skin test) within 14 days prior to randomization
* Patient must have chest computed tomography (CT) scan without contrast performed =< 14 days before randomization. Patient must not have a contraindication for CT

Exclusion Criteria:

* Patient must not have clinical evidence of cardiac dysfunction (as determined by the treating investigator) as an alternative diagnosis to steroid-refractory pneumonitis
* Patient must not be receiving anti-PD-1/-PD-L1 agent in combination with any of the following anti-cancer agents: docetaxel, cyclophosphamide, gefitinib, erlotinib, osimertinib, crizotinib, bleomycin, afatinib
* Patient must not be receiving concurrent radiation therapy to the chest
* Patient must not be deemed to have radiation pneumonitis. Patients with a history of stable radiation pneumonitis not requiring corticosteroid therapy within the last 3 months prior to randomization will be allowed on study
* Patient must not have pre-existing interstitial lung disease or pneumonitis requiring corticosteroid therapy from any other cause, as determined by the treating investigator
* Patient must not have an absolute contraindication to IVIG or infliximab, including: clinical history of severe hypersensitivity reaction, selective IgA deficiency, active hepatitis B, active tuberculosis, active human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS) where a study subject has a CD4 count of =< 200 at screening, or drug interaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jarushka Naidoo, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (18):
- United States (18):
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Bronson Battle Creek, Battle Creek, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Derived] Beattie J, Rizvi H, Fuentes P, Luo J, Schoenfeld A, Lin IH, Postow M, Callahan M, Voss MH, Shah NJ, Betof Warner A, Chawla M, Hellmann MD. Success and failure of additional immune modulators in steroid-refractory/resistant pneumonitis related to immune checkpoint blockade. J Immunother Cancer. 2021 Feb;9(2):e001884. doi: 10.1136/jitc-2020-001884. PMID 33568350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on June 25, 2020 and one patient was enrolled on January 7, 2021. Due to slow accrual, the study was closed on December 14, 2023.
Period: Overall Study
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one patient was enrolled on this study. Due to the concern on confidentiality, individual data is not reported due to confidentiality reasons.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Pneumonitis Response Rate
Description: Pneumonitis response will be defined as an improvement in partial pressure of arterial oxygen (PaO2)/fraction of inspired oxygen (FiO2) of >= 20% measured by PaO2 and recording of the FiO2 received by the patient at the time of the arterial blood gas assessment, on day 28 compared with day 1.
Time Frame: At day 28
Population: Only one patient was enrolled on this study. Due to confidentiality reasons, individual data was not reported.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Patients With Radiologic Response for Steroid-refractory Pneumonitis
Description: Radiologic features of steroid-refractory pneumonitis will be assessed by percentage lung parenchyma involved, percentage of ground-glass opacity in lung parenchyma, and lung volume on computed tomography. The pneumonitis and lung volume will be graded "Definitely decreased", "Probably decreased", "No significant change", "Probably increased" and "Definitely increased". Response to study therapy will be defined by combining the categories "Definitely decreased" and "Probably decreased".
Time Frame: At days 1, 14, and 28
Population: Only one patient was enrolled so individual data won't be reported due to confidentiality reasons.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Functional Parameters of Steroid-refractory Pneumonitis by Spirometry
Description: Functional features of pneumonitis will be assessed by spirometry (forced vital capacity, forced expiratory volume in one second). These quantitative measures will be reported descriptively (by median, mean, and range) by timepoints and treatment arms.
Time Frame: At days 1, 14, and 28
Population: Only one patient was enrolled, so individual data won't be reported due to confidentiality reasons.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Functional Parameters of Steroid-refractory Pneumonitis by Diffusion Capacity
Description: Functional features of pneumonitis will be assessed by diffusion capacity of the lung. These quantitative measures will be reported descriptively (by median, mean, and range) by timepoints and treatment arms.
Time Frame: At days 1, 14, and 28
Population: Only one patient was enrolled so individual data won't be reported due to confidentiality reasons.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Functional Parameters of Steroid-refractory Pneumonitis by Oxygen Saturation
Description: Functional features of pneumonitis will be assessed by oxygen saturation on room air at rest, collected as part of the vital signs. These quantitative measures will be reported descriptively (by median, mean, and range) by timepoints and treatment arms.
Time Frame: At days 1, 14, and 28
Population: Only one patient was enrolled so individual data won't be reported due to confidentiality reasons.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Deaths Within 28 Days
Description: Death reported in the 28-day period will be tabulated by treatment arm, and classified as pneumonitis-related, immunosuppression related, disease-related or other.
Time Frame: Up to 28 days
Population: Only one patient was enrolled so individual data won't be reported due to confidentiality reasons.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Adverse Events
Description: Will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The number and severity of treatment-related adverse events from infections in any organ system by the CTCAE reported in the 28-day period after additional immunosuppression.
Time Frame: Up to 28 days
Population: Only one patient was enrolled so individual data won't be reported due to confidentiality reasons.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Total Score of Functional Assessment of Cancer Therapy - Lung Version 4
Description: Patient-reported outcomes of steroid-refractory pneumonitis will be measured by questionnaires (Functional Assessment of Cancer Therapy - Lung version 4 [FACT-L]). FACT-L consists of 5 subscales and the total score is calculated by summing the scores of the 36 items. The score ranges between 0 and 136. The higher the score, the better the quality of life.
Time Frame: At days 1, 14, and 28
Population: Only one patient was enrolled, so individual data won't be reported due to confidentiality reasons.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Distribution of Biomarkers in Patients Who Develop Steroid-refractory Pneumonitis
Description: Potential blood/serum biomarkers for pneumonitis will be assessed from serially collected blood/serum in accrued patients (on Days 1, 14 and 28 after study treatment) and controls, whose blood/serum will be obtained as part of a parallel tissue-collection protocol.
Time Frame: Days 1, 14 and 28 after study treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: To Evaluate Associations Between Pneumonitis and Autoantibodies, T Cell Expansion, and Baseline Cytokines in the Blood
Description: To evaluate associations between pneumonitis and autoantibodies, T cell expansion, and baseline cytokines in the blood.
Time Frame: On days 1, 14, and 28 post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks until 30 days after treatment completion, up to 3 years
Description: Only one patient was enrolled on this study. Due to the concern on confidentiality, individual data was not reported.
Arm/Group | Arm A (Infliximab) | Arm B (Intravenous Immunoglobulin Therapy)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Only one patient was enrolled on this study. Due to the concern on confidentiality, individual data was not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT04438382/Prot_SAP_000.pdf